CLINICAL TRIAL: NCT04770402
Title: Acupuncture for Chemo-Induced Peripheral Neuropathy (CIPN) in Multiple Myeloma (MM) Patients- A Randomized Controlled Trial
Brief Title: Acupuncture for Chemo-Induced Peripheral Neuropathy in Multiple Myeloma Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accrual
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Atrium Health Levine Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00081364; 00049444 (Other: Advarra IRB); LCI-SUPP-MYE-ACUP-001 (Other: Atrium Health)
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Results first posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-12

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
Keywords: Neuropathy; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Experimental): Subjects on this arm will receive 12 sessions of acupuncture over approximately 10 weeks, along with continued standard treatment by their physician.
  Interventions: Other: Acupuncture
- Standard of Care (Active Comparator): Subjects on this arm will not receive acupuncture, but will continue to be followed by their physician with standard treatment for their neuropathy.
  Interventions: Other: Standard of Care CIPN management

INTERVENTIONS:
Other: Acupuncture — 12 acupuncture sessions over 10 weeks
  Arms: Acupuncture
Other: Standard of Care CIPN management — Investigator directed standard of care management of CIPN
  Arms: Standard of Care

SUMMARY:
This randomized, controlled trial is designed to evaluate the effect of acupuncture on Chemotherapy-Induced Peripheral Neuropathy (CIPN), other symptoms, and potential opioid and concomitant medication sparing effects in comparison to standard of care management in Multiple Myeloma subjects.

DETAILED DESCRIPTION:
This study aims to strengthen the care of persons with Multiple Myeloma by improving quality of life (QOL) and ability to perform daily activities through reduced Chemotherapy-Induced Peripheral Neuropathy (CIPN) symptoms. CIPN debilitates and erodes QOL by preventing individuals from pursuing their normal activities of daily living.

The features of CIPN, including physical, social/family, emotional, functional, and specific CIPN symptoms, will be measured with the validated FACT-GOG-NTX. This project brings necessary attention and scientific inquiry to supportive cancer care, which is sometimes de-prioritized behind disease treatment. The potential for nonpharmacologic acupuncture to reduce CIPN and other symptoms with minimal side effects has beneficial implications for disease treatment. Patients with controlled symptoms are better able to tolerate life-prolonging treatment and avoid chemotherapy dose reductions which result from neurotoxic side effects of chemotherapy.

Subjects who consent and are determined to be eligible will be randomized to receive either acupuncture treatment or standard of care treatment for their CIPN. Subjects' socio-demographics, medical history, opioid and concomitant medication intake information will be collected. Subjects who are randomized to the acupuncture treatment arm will receive 12 sessions of acupuncture over approximately 10 weeks. Subjects randomized to standard of care will continue with standard of care therapy per their physician for treatment of their CIPN. All subjects will complete questionnaires at Baseline, mid-point, and endpoint. Responses to questionnaires will then be analyzed towards answering the study's objectives.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and HIPAA authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
2. Age ≥ 18 years at the time of consent
3. Subject has diagnosis of Multiple Myeloma (any stage) per Investigator
4. Currently being treated with bortezomib or bortezomib-combination chemotherapy
5. ECOG Performance status of 0-3
6. Life expectancy of ≥ 12 weeks
7. Chemotherapy-Induced Peripheral Neuropathy score of ≥ 2
8. No planned hospital admission in the next 10 weeks
9. As determined by the enrolling physician, ability of the subject to understand and comply with study procedures for the entire length of the study

Exclusion Criteria:

1. Uncontrolled intercurrent illness/medical condition or psychiatric illness/social situations that would limit compliance with study requirements as determined by the investigator
2. Subjects with neuropathy pain as a result of spinal injury or vertebral compression fractures
3. Subjects with needle phobia
4. Previous diagnosis of amyloidosis or POEMS syndrome
5. Local infection at or near the planned acupuncture sites (see Appendix A)
6. Subjects with metastatic involvement of the nervous system/active central nervous system disease
7. Plan to receive Healing Touch or Oncology Massage during study
8. Have received acupuncture within 30 days prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shamille Hariharan, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Levine Cancer Institute, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Acupuncture | Standard of Care
Started | 8 | 4
Completed | 6 | 1
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Non-compliance | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acupuncture | Standard of Care | Total
Number analyzed (Participants) | 8 | 4 | 12
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63.5 [58.5 to 69.5] | 58.0 [56.0 to 68.5] | 62.0 [56.0 to 69.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 7 | 4 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 4 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 4 | 2 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 4 | 12
Baseline Chemotherapy-Induced Peripheral Neuropathy Score [Count of Participants; unit: Participants] — Neuropathy is subject reported using an 11-point scale from 0-no neuropathy to 10-worst possible neuropathy.
  Participants
    4 | 0 | 2 | 2
    5 | 0 | 0 | 0
    6 | 4 | 0 | 4
    7 | 2 | 1 | 3
    8 | 2 | 0 | 2
    9 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change of Neuropathy in Actively Treated Multiple Myeloma Subjects Diagnosed With Chemotherapy-induced Peripheral Neuropathy Who Received Acupuncture vs Standard of Care Management.
Description: Neuropathy will be subject reported using an 11-point scale from 0-no neuropathy to 10-worst possible neuropathy. The outcome will be measured as a binary variable indicating whether or not a subject experienced at least a 2-point improvement in neuropathy between the baseline score and the score obtained at Week 10 +/- 1 week.
Time Frame: Approximately 10 weeks, from baseline measure to 10 week (+/- 1 week) measure.
Population: The analysis population are those that met the evaluable population criteria, which was enrolled subjects who have complete baseline and Week 10 neuropathy scores.
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Standard of Care
Number analyzed (Participants) | 7 | 1
Participants
  Experienced at least a 2 point improvement in neuropathy between baseline and Week 10 | 6 | 0
  Did not experience at least a 2 point improvement in neuropathy between baseline and Week 10 | 1 | 1

2. Secondary Outcome: Specific Features of Chemotherapy-Induced Peripheral Neuropathy From FACT-GOG-NTX
Description: Specific features of CIPN assessed through the subscale from FACT-GOG-NTX will be determined for each subject as a composite measure, which is calculated as the sum of the responses to the subscale questions. For subjects who complete all 12 subscale questions, the composite score will range from 0 to 48. Higher scores mean worse outcome
Time Frame: 10 weeks
Population: as for outcome 1
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | Acupuncture | Standard of Care
Number analyzed (Participants) | 7 | 1
Score on a scale | 14.0 [5.0 to 27.0] | 23.0 [23.0 to 23.0]

3. Secondary Outcome: Nausea - FACT-GOG-NTX
Description: Nausea will be determined for each subject as 5 level ordinal variable from 0 = not at all to 4 = very much through question GP2 on the FACT-GOG-NTX subject-reported assessment. The item is to rate the statement 'I have nausea.'
Time Frame: approx. 10 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Standard of Care
Number analyzed (Participants) | 7 | 1
Participants
  Not at all | 7 | 1
  A little bit | 0 | 0
  Somewhat | 0 | 0
  Quite a bit | 0 | 0
  Very much | 0 | 0

4. Secondary Outcome: Sadness- FACT-GOG-NTX
Description: Sadness will be determined for each subject as 5 level ordinal variable from 0 = not at all to 4 = very much through question GE1 on the FACT-GOG-NTX subject-reported assessment. The item is to rate the statement 'I feel sad'.
Time Frame: approx. 10 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Standard of Care
Number analyzed (Participants) | 7 | 1
Participants
  Not at all | 4 | 1
  A little bit | 2 | 0
  Somewhat | 1 | 0
  Quite a bit | 0 | 0
  Very much | 0 | 0

5. Secondary Outcome: Nervousness- FACT-GOG-NTX
Description: Nervousness will be determined for each subject as 5 level ordinal variable from 0 = not at all to 4 = very much through question GE4 on the FACT-GOG-NTX subject-reported assessment. The item is to rate the statement 'I feel nervous.'
Time Frame: approx. 10 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Standard of Care
Number analyzed (Participants) | 7 | 1
Participants
  Not at all | 4 | 1
  A little bit | 3 | 0
  Somewhat | 0 | 0
  Quite a bit | 0 | 0
  Very much | 0 | 0

6. Secondary Outcome: Sleep Quality- FACT-GOG-NTX
Description: Sleep quality will be determined for each subject as 5 level ordinal variable from 0 = not at all to 4 = very much through question GF5 on the FACT-GOG-NTX subject-reported assessment. The item is to rate the statement 'I am sleeping well.'
Time Frame: approx. 10 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Standard of Care
Number analyzed (Participants) | 7 | 1
Participants
  Not at all | 0 | 0
  A little bit | 0 | 0
  Somewhat | 4 | 0
  Quite a bit | 2 | 0
  Very much | 1 | 1

7. Secondary Outcome: Lack of Energy- FACT-GOG-NTX
Description: Lack of energy will be determined for each subject as 5 level ordinal variable from 0 = not at all to 4 = very much through question GP1 on the FACT-GOG-NTX subject-reported assessment. The item is to rate the statement 'I have a lack of energy.'
Time Frame: approx. 10 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Standard of Care
Number analyzed (Participants) | 7 | 1
Participants
  Not at all | 2 | 0
  A little bit | 3 | 0
  Somewhat | 2 | 1
  Quite a bit | 0 | 0
  Very much | 0 | 0

8. Secondary Outcome: Pain- FACT-GOG-NTX
Description: Pain will be determined for each subject as 5 level ordinal variable from 0 = not at all to 4 = very much through question GP4 on the FACT-GOG-NTX subject-reported assessment. The item is to rate the statement 'I have pain.'
Time Frame: approx. 10 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Standard of Care
Number analyzed (Participants) | 7 | 1
Participants
  Not at all | 1 | 0
  Very little | 3 | 0
  Somewhat | 2 | 0
  Quite a bit | 1 | 1
  Very much | 0 | 0

9. Secondary Outcome: Constipation
Description: Constipation will be determined for each subject as a 5-level ordinal variable from 0 = not at all to 4 = very much through additional question amended to FACT-GOG-NTX subject-reported assessment. The item is to rate the statement 'I have constipation.'
Time Frame: approx. 10 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Standard of Care
Number analyzed (Participants) | 7 | 1
Participants
  Not at all | 0 | 0
  A little bit | 5 | 0
  Somewhat | 1 | 1
  Quite a bit | 1 | 0
  Very much | 0 | 0

10. Secondary Outcome: Dizziness
Description: Dizziness will be determined for each subject as a 5- level ordinal variable from 0 = not at all to 4 = very much through additional question amended to FACT-GOG-NTX subject-reported assessment. This item is to rate the statement 'I have dizziness'.
Time Frame: approx. 10 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Standard of Care
Number analyzed (Participants) | 7 | 1
Participants
  Not at all | 1 | 0
  A little bit | 3 | 1
  Somewhat | 2 | 0
  Quite a bit | 1 | 0
  Very much | 0 | 0

11. Secondary Outcome: Dry Mouth
Description: Dry mouth will be determined for each subject as a 5- level ordinal variable from 0 = not at all to 4 = very much through additional question amended to FACT-GOG-NTX subject-reported assessment. This item is to rate the statement 'I have dry mouth.'
Time Frame: approx. 10 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Standard of Care
Number analyzed (Participants) | 7 | 1
Participants
  Not at all | 1 | 0
  A little bit | 5 | 0
  Somewhat | 0 | 1
  Quite a bit | 1 | 0
  Very much | 0 | 0

12. Secondary Outcome: General Health - CDC-HRQOL
Description: General Health assessed through CDC-HRQOL Question 1 will be calculated for each subject as a 5- level ordinal variable from Poor to Excellent.
Time Frame: approx. 10 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Standard of Care
Number analyzed (Participants) | 7 | 1
Participants
  Excellent | 0 | 0
  Very good | 1 | 0
  Good | 4 | 1
  Fair | 2 | 0
  Poor | 0 | 0

13. Other Pre Specified Outcome: Adverse Events of Special Interest
Description: Adverse Events of Special Interest (AESI) will be determined for each subject as binary variables indicating whether or not they experienced a protocol defined AESI, including bleeding, bruising, skin infection, edema, dry skin, urticaria, pruritus, rash, pain or flushing at the acupuncture site, or dizziness, syncope, fatigue, or hyperhidrosis.
Time Frame: approx. 10 weeks
Population: Enrolled participants on the acupuncture arm
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Standard of Care
Number analyzed (Participants) | 7 | 0
Participants | 0 |

14. Other Pre Specified Outcome: Opioid Use
Description: Opioid use will be calculated for each subject as a quantitative value assessed through Morphine Equivalent Daily Dose (MEDD).
Time Frame: approx. 10 weeks
Population: All participants receiving acupuncture or standard of care
Measure: Median (Full Range); unit: morphine milligram equivalents per day
Arm/Group | Acupuncture | Standard of Care
Number analyzed (Participants) | 7 | 4
morphine milligram equivalents per day | 0.0 [0.0 to 0.0] | 82.5 [15.0 to 150.0]

15. Other Pre Specified Outcome: Acupuncture Administration
Description: Acupuncture administration will be defined for each subject on the acupuncture arm as the number of attended acupuncture sessions from 0 to 12.
Time Frame: approx. 10 weeks
Population: Enrolled participants randomized to the acupuncture arm
Measure: Median (Full Range); unit: number of acupuncture sessions
Arm/Group | Acupuncture | Standard of Care
Number analyzed (Participants) | 7 | 0
number of acupuncture sessions | 11 [9 to 12] |

16. Other Pre Specified Outcome: Acupuncture Expectancy
Description: The acupuncture expectancy score will be captured quantitatively for each subject as a composite score ranging from 4 to 20. Higher scores indicate higher expectancy of acupuncture.
Time Frame: approx 10 weeks
Population: Participants randomized to the acupuncture arm
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | Acupuncture | Standard of Care
Number analyzed (Participants) | 8 | 0
Score on a scale | 13 [7 to 20] |

ADVERSE EVENTS:
Time Frame: AESIs were collected for approximately 10 weeks for the duration of the acupuncture treatment (for those on the intervention arm) and collected through 30 days after last acupuncture session. Serious adverse events and all-cause mortality were monitored and collected for both arms throughout the study, approximately 10 weeks.
Description: Only All-Cause Mortality, Serious Adverse Events, and Adverse Events of Special Interest (AESI) were collected for this study. All-cause mortality and Serious Adverse Events were collected for both arms as defined in the clinicaltrials.gov definition. AESIs were collected only for subjects on the intervention arm, including bleeding, bruising, skin infection, edema, dry skin, urticaria, pruritus, rash, pain or flushing at the acupuncture site, dizziness, syncope, fatigue, or hyperhidrosis.
Arm/Group | Acupuncture | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/4
Other Adverse Events (participants affected / at risk) | 0/8 | 0/0

LIMITATIONS AND CAVEATS:
Early termination due to low accrual leading to small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-21): https://cdn.clinicaltrials.gov/large-docs/02/NCT04770402/Prot_SAP_001.pdf
  • Informed Consent Form (2023-04-13): https://cdn.clinicaltrials.gov/large-docs/02/NCT04770402/ICF_000.pdf